CLINICAL TRIAL: NCT06023706
Title: Phase 3 Confirmatory, Randomised 1:1 Double-blind, Placebo-controlled Study Evaluating the Analgesic Efficacy of Capsaicin 8% Patches in Chronic Coccygodynia.
Brief Title: Study Evaluating the Analgesic Efficacy of Capsaicin 8% Patches in Chronic Coccygodynia.
Acronym: CAPSACOX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC22_0415
Record Dates: First submitted 2023-08-01; First posted 2023-09-05 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Coccyx Disorder; Neuropathic Pain; Coccygodynia
MeSH Terms: conditions — Neuralgia | interventions — Capsaicin; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capsaicin 179 mg cutaneous patch (Experimental): Capsaicin 179 mg cutaneous patch.
  1 patch applied once for 1 hour at inclusion visit.
  Interventions: Drug: Capsaicin 179 Mg Cutaneous Patch
- Capsaicin low concentration patch (Placebo Comparator): Capsaicin 0.04 cutaneous patch.
  1 patch applied once for 1 hour at inclusion visit
  Interventions: Drug: Capsaicin low concentration patch (capsaicin 0,04%, 3,2 mg/cm2)

INTERVENTIONS:
Drug: Capsaicin 179 Mg Cutaneous Patch — 1 patch applied once for 1 hour
  Other Names: qutenza
  Arms: Capsaicin 179 mg cutaneous patch
Drug: Capsaicin low concentration patch (capsaicin 0,04%, 3,2 mg/cm2) — 1 patch applied once for 1 hour
  Arms: Capsaicin low concentration patch

SUMMARY:
The primary objective is to demonstrate the analgesic effect at day 60 of 8% capsaicin patch (Qutenza) for the treatment of patients with coccygodyinia.

DETAILED DESCRIPTION:
This trial is a French, multicenter, randomized, controlled, bouble-blind and prospective study. Patients enrolled will be clinically followed for 5 months. The treatment duration per subject is 1 hour (1time).

ELIGIBILITY:
Inclusion Criteria:

* >18 years old at the pre-inclusion visit
* Presenting with chronic coccygodynia: pain in the coccygeal region, increased by sitting and or when rising from a sitting position and pain over the last ten days of intensity greater than or equal to four on the eleven-point numerical scale (from zero to ten) and having been present for more than 3 months.
* Failure of previous treatments: NSAIDs, pressure-relieving cushions and/or infiltration or having a contraindication to these treatments, or not wishing to receive these treatments
* Have never been treated with an 8% capsaicin patch for this indication
* With at least one clinical sign suggestive of neuropathic pain (burning, painful cold, numbness, tingling, electric discharge, allodynia of the gluteal groove, allodynia to pressure on the coccyx)
* Proficiency in reading and writing the French language
* Be affiliated to the social security system
* Have signed an informed consent form
* Women must meet one of the following criteria at the time of inclusion:
* be using adequate contraceptive measures, and have a negative pregnancy test (specify if urine or blood test) prior to receiving the first dose of trial medication;
* or be post-menopausal (aged over 50 with amenorrhoea for at least 12 months after stopping all exogenous hormonal treatments)
* or (if under 50) have been in amenorrhoea for at least 12 months after stopping all exogenous hormone treatments and with luteinising hormone (LH) and follicle stimulating hormone (FSH) levels corresponding to post-menopausal levels.
* or have undergone irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy (this operation must be documented).

Exclusion Criteria:

* Coccygodynia accompanied by a dermatological lesion in the intergluteal cleft (psoriasis, pilodinial cyste, wound)
* Patients with other major pain disorders likely to interfere with pain assessment
* Hypersensitivity to capsaicin or to one of the excipients
* Adults under legal protection (guardianship, curatorship, legal protection)
* Pregnant or breast-feeding women
* Patients who have undergone total coccygectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
to demonstrate the analgesic effect at day 60 of 8% capsaicin patch (Qutenza) for the treatment of patients with coccygodyinia. | Day 60
  The difference in the proportion of subjects improved (PGIC≤2) in either treatment group at day 60. It is expected that there will be a difference of at least 20% between treatment arms.

SECONDARY OUTCOMES:
Evaluation of the tolerability of the 8% capsaicin patch compared to low concentration capsaicin patch (control) within the first 7 days | time 0 (prior to patch application), hour 1, 6, 12, 24, day 2 and day 7 and by collecting AEs during the study.time 0 (prior to patch application), hour 1, 6, 12, 24, day 2 and day 7 and through study completion (an average of 5 months)
  Tolerability will be assessed by the evolution over time of the pain intensity in standing position in the treated zone as measured on an 11 point numeric rating scale at time 0 (prior to patch application), hour 1, 6, 12, 24, day 2 and day 7 and by collecting AEs during the study.
Evaluate the safety of the capsaicin 8% patch compared with the control patch throughout the study. | Throughout the study (an average of 5 months)
  Safety will be assessed by recording and describing adverse events throughout the study.
Evaluation of the analgesic effect over time and maintenance of effect in the two treatment groups over the entire study. | Day 2, Day 7, Day 15, Day 21, Day 30, Day 45, Day 60, Day 90, Day 120 and Day 150.
  The timecourse of the analgesic effect will be measured by the Patients' Global Impression of Change (PGIC) scale and the area under the pain intensity score in sitting position as measured Day 2, Day 7, Day 15, Day 21, Day 30, Day 45, Day 60, Day 90, Day 120 and Day 150.
Evaluation of health care consumption in the two treatment groups over the entire study period (5 months). | Over 5 months
  Care consumption will be assessed over 5 months using the Medication Quantification Scale (MQS), which provides a standardised assessment of consumption of analgesics and co-antalgesics.
Evaluation of health care consumption in the two treatment groups over the entire study period (5 months). | Over 5 months
  Care consumption will be assessed over 5 months using a self-diary in which patients will enter the dates of medical consultations (psychiatry, rheumatology, general medicine, etc.), para-medical consultations and/or complementary medical consultations (physiotherapy, acupuncture, osteopathy, psychotherapy, etc.).
Evaluation of the cost-utility of 8% capasaicin patch with common clinical practice over a time horizon of 5 months | Over a time horizon of 5 months
  The evaluation of cost-utility will be assessed as the ratio of the incremental cost-utility (RICU in cost per QALY gained) comparing the treatment with 8% capsaicin patch with usual practice according to the collective perspective and a 5-month horizon. QALYS will be calculated using patients' lifespan and a utility score obtained from responses to the EQ-5D-5L generic quality of life questionnaire.
Analysis of primary and secondary endpoints according to the presence or absence of sacrococcygeal hypermobility. | At inclusion
  Subgroup analysis according to the presence or absence of a sacrococcygeal mobility disorder at inclusion for the primary endpoint and the first two secondary endpoints.
Determination of the therapeutic response to 8% capsaicin patch | Day 60
  Measurement of the association between the patient's intrinsic clinical parameters and a therapeutic response to capsaicin defined by a PGIC ≤2.
Sensitivity study to compare results on the primary endpoint by comparing data from the PGI-C and a comparison of the two numerical pain assessments at Day 0 and Day 60. | Between Day 0 and Day 60
  Comparison of the classification of patients as success-failure between PGI-C values at Day 60 (success if PGI-C≤2) and numerical pain assessments between Day 0 and Day 60 (success if there is a reduction of at least 2 points on the EN).

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Brest University Hospital, Brest
  - Vendée Departmental Hospital, La Roche-sur-Yon
  - Confluent Private Hospital Centre, Nantes
  - Nantes University Hospital, Nantes
  - GH Paris saint Joseph, Paris
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: Undecided